CLINICAL TRIAL: NCT06842316
Title: In Vitro Effects of Phytocannabinoids on Immune Response and Autophagy During Chronic Immune-mediated Inflammatory Diseases
Brief Title: Effects of Phytocannabinoids on Immune Response and Autophagy During Chronic Immune-mediated Inflammatory Diseases
Acronym: pCB-IMIDs
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHUO-2024-14
Record Dates: First submitted 2025-02-13; First posted 2025-02-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Disorder of Immune System; Spondylitis, Ankylosing; Arthritis, Rheumatoid; Arthritis, Psoriatic; Inflammatory Bowel Diseases; Sjogren's Syndrome; Lupus Erythematosus, Systemic
Keywords: IMIDs; phytocanabinoid; inflammatory effect; blood cells
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Rheumatoid; Arthritis, Psoriatic; Inflammatory Bowel Diseases; Sjogren's Syndrome; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample : 40 ml of blood corresponding to 1 tube EDTA of 10 ml and 3 heparinized tubes for RNA analyzes, Multiplexed ELISA and in vitro stimulations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Rheumatoid polyarthritis: 10 patients without, 10 patients under basic treatment (csDMARDs*) and 10 patients under biotherapy or targeted therapy
  Interventions: Other: 1 blood sample, 40 mL (collection during a blood test, part of the standard of care for this disease)
- Spondyloarthropathy: 20 patients with or without IBD, including 10 under biotherapy or targeted therapy
  Interventions: Other: 1 blood sample, 40 mL (collection during a blood test, part of the standard of care for this disease)
- Psoriatic arthritis: 10 patients without, 10 patients with basic treatment (csDMARD) and 10 patients under biotherapy or targeted therapy
  Interventions: Other: 1 blood sample, 40 mL (collection during a blood test, part of the standard of care for this disease)
- Systemic lupus erythematosus: 10 patients with connective tissue disease (Systemic lupus erythematosus)
  Interventions: Other: 1 blood sample, 40 mL (collection during a blood test, part of the standard of care for this disease)
- Sjögren's syndrome: 10 patients with connective tissue disease (Sjögren's syndrome)
  Interventions: Other: 1 blood sample, 40 mL (collection during a blood test, part of the standard of care for this disease)

INTERVENTIONS:
Other: 1 blood sample, 40 mL (collection during a blood test, part of the standard of care for this disease) — Mononuclear and polynuclear peripheral blood cells from subjects suffering from IMID will be exposed in vitro to different inflammatory inducers with and without the concomitant addition of at least 4 different pCB extracts spectrum complete (full spectrum) including a dominant CBD extract and low in THC (<0.2%), 1 dominant THC extract, 1 balanced THC/CBD extract and 1 dominant CBG extract. The same analyzes will be carried out in the presence of a recognized anti-inflammatory (for example hydrocortisone or dexamethasone) which will thus be used as a positive control.

SUMMARY:
Cannabis, in addition to its psychotropic properties, could have anti-inflammatory and immunomodulatory effects. Phytocannabinoids (pCBs) are a group of molecules naturally secreted by the cannabis plant. The major pCBs are cannabidiol (CBD) and Δ9-tetrahydrocannabinol Δ9 (THC). Only THC has psychotropic effects, which CBD does not have. Alongside these two main components, there is a wide variety of other molecules, such as other pCBs and terpenes which could increase the effects on immune system through synergistic interactions between these different compounds ("entourage effect").In vivo, pCBs essentially interfere with the endocannabinoid system, acting on many ubiquitous receptors, present on a significant number of different cell types. Numerous published studies show that pCBs have immunomodulatory and anti-inflammatory properties by acting on several of these receptors, whether through modulation of the immune response of different cell types, effects on cytokine networks, reduction of innate and adaptive responses and/or impact on cell survival or death (autophagy, proliferation/ apoptosis). The Immune-Mediated Inflammatory Diseases (IMIDs) affect 5 to 7% of the general population in Western countries, involve different organs (joints, skin, digestive tract) but share the same inflammatory mechanisms resulting from a dysregulation of the immune response. Our research focuses on the identification of the most effective phytochemical profile of pCBs, allowing an optimal effect on chronic inflammatory pathologies of interest among immune-mediated chronic inflammatory diseases (IMIDs). The pCB-IMIDs project is therefore part of an innovative translational project, around new therapeutic applications of medical cannabis (CannAppIMIDs). In our study, we will include 100 patients with one of IMIDs among Rheumatoid Arthritis, spondylarthritis, psoriatic arthritis, Sjogren disease and systemic lupus, at different stage and with different treatments. After patient's consent we will collect for research purposes an additional 40 ml of blood during a routine care blood test. Mononuclear and polynucleated blood cells will be exposed in vitro to different full-spectrum pCB extracts (full spectrum extract) including a CBD dominant and low THC extract (<0.2%), 1 dominant THC extract, 1 balanced THC/CBD extract and 1 dominant CBG extract. In this cross-sectional study, our objective will be to assess the biological effects of different pCB compositions on inflammatory profiles (concentrations of pro and anti-inflammatory cytokines and chemokines) and modulations of expression profiles (autophagy, apoptosis, and cannabinoid receptor expression profile).

DETAILED DESCRIPTION:
Background:

The analgesic and anxiolytic properties of cannabis are at the origin of the French experiment on medical cannabis set up in 2020 and led by the ANSM (National Agency for the Safety of Medicines and Health Products) for 5 well-identified pathologies (neuropathic pain, certain forms of pediatric epilepsy, symptoms linked to cancer or anti-cancer treatment, palliative situations and painful spasticity linked to multiple sclerosis). Phytocannabinoids (pCBs) are a group of molecules naturally secreted by the cannabis plant. The main pCBs are cannabidiol (CBD) and Δ9-tetrahydrocannabinol Δ9-THC [1, 2]. Only THC has psychotropic effects, which CBD does not have. Alongside these two main components, there is a wide variety of molecules [cannabigerol (CBG), cannabinol (CBN), cannabichromene (CBC) and other terpenes] which are said to have an "entourage effect" by increasing the effects by synergistic interactions between these different compounds [3-7]. CBD of natural origin can be purified without other terpenes corresponding to CBD alone ("CBD isolate") or is combined with terpenes and phytocannabinoids but without THC or any other pCB ("broad spectrum"), or in unpurified form, CBD with terpenes and THC ("full spectrum").

In vivo, pCBs essentially interfere with the endocannabinoid system, acting on numerous receptors present on a large number of different cell types [8]. This means that pCBs can be used to treat a wide range of organs. Numerous published works show that pCBs have immunomodulatory and anti-inflammatory properties by acting on several of these receptors, whether via modulation of the immune response of different cell types, effects on cytokine networks, reduction of innate and adaptive responses [9, 10] and/or impact on cell survival or death (autophagy, proliferation/apoptosis) [8, 9]. Thus, in addition to its neurological effects [10, 11], cannabis possesses anti-inflammatory, pro-autophagic and anti-proliferative properties, which are still imperfectly characterized.

Understanding the mechanisms of action of pCBs, individually or in combination with other molecules present in cannabis, on different therapeutic targets therefore presents an immense challenge in the management of Immune-Mediated Inflammatory Diseases (IMIDs). These IMIDs affect 5 to 7% of the general population in Western countries, and involve different organs (joints, skin, gut) but share the same inflammatory mechanisms, resulting from a deregulation of the immune response.

The pCB-IMIDs project is part of an innovative translational project focusing on new therapeutic applications for medical cannabis (CannAppIMIDs).

Objectives:

The objective of this exploratory project is to evaluate the biological and immunological effects of exposure of blood cells from patients suffering from IMID to different varieties of pCB extracts on:

1. The inflammatory profile (main objective)
2. The expression profile of cannabinoid receptors
3. The autophagic and apoptotic profile

Methods: Single-center cross-sectional study without prospective follow-up of participants, classified non-interventional study. The study consists, after obtaining consent and verifying the eligibility criteria (with saliva test specific to the study), in taking an additional 40 ml of blood during a planned blood test for research purposes and to collect medical data on patients and their inflammatory pathology.

Mononuclear and polynuclear blood cells from subjects suffering from IMID will be exposed in vitro to different inflammatory inducers used individually and/ or all together (LPS- bacterial Lipopolysaccahride, TLR-4 ligand and/or poly-I:C , TLR-3 ligand and/or PAM3CSK4, TLR1/TLR2 ligand, and/or PHA-P - phytohemagglutin P, polysaccharide and glycoprotein ligand) with and without the concomitant addition of different complete spectrum of pCB extracts (full spectrum) including a dominant CBD extract and low in THC (<0.2%), 1 dominant THC extract, 1 balanced THC/CBD extract and 1 dominant CBG extract. The same analyzes will be carried out in the presence of a recognized anti-inflammatory (for example hydrocortisone or dexamethasone) which will thus serve as a positive control [12].

All analyses will be carried out at CBM - UPR4301 CNRS. Results will allow us to formulate hypotheses, guide and argue for future clinical research studies evaluating the benefit(s) and tolerance of extracts rich in pCB in taking in therapeutic management of IMIDs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old
2. Diagnosis confirmed by a rheumatologist of RA or spondyloarthropathy (with or without IBD) or psoriatic arthritis (with or without active psoriasis) or systemic lupus erythematosus or Sjögren's disease
3. Patient who has expressed consent to participate in the study
4. Patients affiliated to social security
5. Treatments authorized as part of routine care: non-steroidal anti-inflammatory drugs (NSAIDs), level 1 to 3 analgesics, local corticosteroids, oral corticosteroid therapy (daily dose ≤15 mg/d), 5-aminosalicylic acid, salazopyrine, methotrexate, leflunomide, hydroxychloroquine, biotherapies and targeted therapies.

Exclusion Criteria:

1. Patient who received intravenous corticosteroid therapy less than 4 weeks ago
2. Patient receiving oral corticosteroid therapy with a daily dose >15 mg/day
3. Consumption of CBD and/or recreational cannabis and/or positive saliva test for cannabis consumption and/or CBD
4. Pregnant and lactating women
5. Persons under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this exploratory study, the study population will include subjects suffering from IMID with rheumatological expression: rheumatoid arthritis (RA), Spondyloarthropathies with or without IBD, Psoriatic arthritis (Rpso), systemic lupus erythematosus (SLE), Sjögren's disease.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2027-04-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to evaluate the biological effect of exposure of blood cells from patients suffering from IMID to different varieties of pCB extracts on the inflammatory profile. | One sample at inclusion for all patients
  The initial inflammatory profiles of patients will be established by evaluations at the transcriptomic and protein level.
The primary outcome is to evaluate the immunological effect of exposure of blood cells from patients suffering from IMID to different varieties of pCB extracts on the inflammatory profile. | One sample at inclusion for all patients
  In plasma, the concentrations of cytokines and chemokines associated with inflammation, pro (mainly TNF-α IFN-α, but for instance also IL6, IL8, and IL1-β) and anti-inflammatory (for example IL-10) will be quantified in Multiplexed (34-plex type) or conventional ELISA. The level of expression of the corresponding transcripts, produced by the sorted subpopulations (cellular targets: polymorphonuclear, CD14+ monocyte, CD19+ B lymphocytes, CD4+ T4 lymphocytes and CD8+ T8 lymphocytes) will subsequently be reported by BRB-Seq [13] and/or by droplet RT-PCR (RT-ddPCR) assays. This quantification technique is reproducible, requires little starting biological material and is very efficient in detecting small quantities.

SECONDARY OUTCOMES:
Inflammatory and autophagic/apoptotic transcripts, as well as transcripts of the main phytocannabinoid receptors in subpopulations of sorted blood cells. | One sample at inclusion for all patients
  Quantify ex vivo (by BRB-Seq and/or droplet quantitative RT-PCR (RT-ddPCR)). nflammatory and autophagic/apoptotic transcripts, as well as transcripts of the main phytocannabinoid receptors in subpopulations of sorted blood cells (polymorphonuclear cells, CD14+ monocytes, CD19+ B lymphocytes, CD4+ T and CD8+ T cells and if possible, quantify the evolution, after induction of an inflammatory context, of transcripts.
The main phytocannabinoid receptors in blood cells | One sample at inclusion for all patients
  Quantify ex vivo (by BRB-Seq and/or droplet quantitative RT-PCR (RT-ddPCR)). the expression profile of phyto and endocannabinoid receptors in the subpopulations will be established. Note that the development of this quantification of the transcripts of certain cytokines and several pCB receptors has already been carried out during previous work in the CBM laboratory (on French blood institution blood donors). Finally, an evaluation of mRNAs associated with apoptosis and autophagy could also be documented. Indeed, autophagy, a crucial biological function for the cell, linked to inflammation [14, 15], will also be evaluated, because the combined effects of pCB, pro-apoptotic, pro-autophagic and anti-inflammatory, have already been reported.
The main autophagy genes and apoptosis genes such as caspases | One sample at inclusion for all patients
  Quantify ex vivo (by BRB-Seq and/or droplet quantitative RT-PCR (RT-ddPCR)). Inflammatory and autophagic/apoptotic transcripts, as well as transcripts of the main phytocannabinoid receptors in subpopulations of sorted blood cells (polymorphonuclear cells, CD14+ monocytes, CD19+ B lymphocytes, CD4+ T and CD8+ T cells, and quantify the evolution, after induction of an inflammatory context, of transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Carine Pr SALLIOT, Principal Investigator — CHU Orléans
Locations (1):
- CHU d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Boychuk DG, Goddard G, Mauro G, Orellana MF. The effectiveness of cannabinoids in the management of chronic nonmalignant neuropathic pain: a systematic review. J Oral Facial Pain Headache. 2015 Winter;29(1):7-14. doi: 10.11607/ofph.1274. PMID 25635955
- [Background] Phillips RS, Friend AJ, Gibson F, Houghton E, Gopaul S, Craig JV, Pizer B. Antiemetic medication for prevention and treatment of chemotherapy-induced nausea and vomiting in childhood. Cochrane Database Syst Rev. 2016 Feb 2;2(2):CD007786. doi: 10.1002/14651858.CD007786.pub3. PMID 26836199
- [Background] MECHOULAM R, GAONI Y. A TOTAL SYNTHESIS OF DL-DELTA-1-TETRAHYDROCANNABINOL, THE ACTIVE CONSTITUENT OF HASHISH. J Am Chem Soc. 1965 Jul 20;87:3273-5. doi: 10.1021/ja01092a065. No abstract available. PMID 14324315
- [Background] Costiniuk CT, Saneei Z, Routy JP, Margolese S, Mandarino E, Singer J, Lebouche B, Cox J, Szabo J, Brouillette MJ, Klein MB, Chomont N, Jenabian MA. Oral cannabinoids in people living with HIV on effective antiretroviral therapy: CTN PT028-study protocol for a pilot randomised trial to assess safety, tolerability and effect on immune activation. BMJ Open. 2019 Jan 17;9(1):e024793. doi: 10.1136/bmjopen-2018-024793. PMID 30659041
- [Background] Hanus LO, Meyer SM, Munoz E, Taglialatela-Scafati O, Appendino G. Phytocannabinoids: a unified critical inventory. Nat Prod Rep. 2016 Nov 23;33(12):1357-1392. doi: 10.1039/c6np00074f. PMID 27722705
- [Background] Russo EB. Taming THC: potential cannabis synergy and phytocannabinoid-terpenoid entourage effects. Br J Pharmacol. 2011 Aug;163(7):1344-64. doi: 10.1111/j.1476-5381.2011.01238.x. PMID 21749363
- [Background] Costa L, Amaral C, Teixeira N, Correia-da-Silva G, Fonseca BM. Cannabinoid-induced autophagy: Protective or death role? Prostaglandins Other Lipid Mediat. 2016 Jan;122:54-63. doi: 10.1016/j.prostaglandins.2015.12.006. Epub 2015 Dec 28. PMID 26732541
- [Background] Koay LC, Rigby RJ, Wright KL. Cannabinoid-induced autophagy regulates suppressor of cytokine signaling-3 in intestinal epithelium. Am J Physiol Gastrointest Liver Physiol. 2014 Jul 15;307(2):G140-8. doi: 10.1152/ajpgi.00317.2013. Epub 2014 May 15. PMID 24833710
- [Background] Lattanzi S, Brigo F, Trinka E, Zaccara G, Cagnetti C, Del Giovane C, Silvestrini M. Efficacy and Safety of Cannabidiol in Epilepsy: A Systematic Review and Meta-Analysis. Drugs. 2018 Nov;78(17):1791-1804. doi: 10.1007/s40265-018-0992-5. PMID 30390221
- [Background] Reddy DS. Therapeutic and clinical foundations of cannabidiol therapy for difficult-to-treat seizures in children and adults with refractory epilepsies. Exp Neurol. 2023 Jan;359:114237. doi: 10.1016/j.expneurol.2022.114237. Epub 2022 Oct 4. PMID 36206806
- [Background] Becker L, Holtmann D. Anti-inflammatory effects of alpha-humulene on the release of pro-inflammatory cytokines in lipopolysaccharide-induced THP-1 cells. Cell Biochem Biophys. 2024 Jun;82(2):839-847. doi: 10.1007/s12013-024-01235-7. Epub 2024 Feb 22. PMID 38388989
- [Background] Alpern D, Gardeux V, Russeil J, Mangeat B, Meireles-Filho ACA, Breysse R, Hacker D, Deplancke B. BRB-seq: ultra-affordable high-throughput transcriptomics enabled by bulk RNA barcoding and sequencing. Genome Biol. 2019 Apr 19;20(1):71. doi: 10.1186/s13059-019-1671-x. PMID 30999927
- [Background] Qian M, Fang X, Wang X. Autophagy and inflammation. Clin Transl Med. 2017 Dec;6(1):24. doi: 10.1186/s40169-017-0154-5. Epub 2017 Jul 26. PMID 28748360
- [Background] Zhong Z, Sanchez-Lopez E, Karin M. Autophagy, Inflammation, and Immunity: A Troika Governing Cancer and Its Treatment. Cell. 2016 Jul 14;166(2):288-298. doi: 10.1016/j.cell.2016.05.051. PMID 27419869
- [Background] Liu QR, Aseer KR, Yao Q, Zhong X, Ghosh P, O'Connell JF, Egan JM. Anti-Inflammatory and Pro-Autophagy Effects of the Cannabinoid Receptor CB2R: Possibility of Modulation in Type 1 Diabetes. Front Pharmacol. 2022 Jan 18;12:809965. doi: 10.3389/fphar.2021.809965. eCollection 2021. PMID 35115945